CLINICAL TRIAL: NCT01637870
Title: Negative Pressure Wound Therapy to Prevent Post Operative Wound Complications Following Cesarean Delivery in Women at High Risk for Wound Complications
Brief Title: Negative Pressure Wound Therapy After Cesarean Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbey Hardy-Fairbanks (Other)
Collaborators: Kinetic Concepts, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Abbey Hardy-Fairbanks, Associate Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 201109727
Record Dates: First submitted 2012-07-06; First posted 2012-07-11 (Estimated); Results first posted 2018-04-18 (Actual); Last update posted 2018-04-18 (Actual); Status verified 2018-03

CONDITIONS: Major Puerperal Infection, Postpartum; Wound Complications; Wound Seroma; Caesarean Section Wound Separation; Wound Infection
Keywords: Cesarean delivery; Postpartum infection; Wound complications; Wound seroma; Wound separation; Wound infection; Negative pressure
MeSH Terms: conditions — Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Negative pressure pump (Experimental): Will have the Prevena negative pressure wound system placed at the time of surgery.
  Interventions: Device: Prevena negative pressure wound system

INTERVENTIONS:
Device: Prevena negative pressure wound system — Placement of negative pressure wound system at the time of cesarean delivery for those at increased risk for wound complication

SUMMARY:
This study is aimed at determining whether or not the use of a wound suction device placed on the cesarean incision instead of a standard sterile dressing will decrease the prevalence of wound complications and wound infections in women at high risk for post operative complications. The study will first look at the infection and wound complication rate in women 6 months prior to the start date of the study by reviewing charts of women who have undergone a cesarean section. The study involves placing a single use, portable wound vacuum over the cesarean section incision and keeping it in place for 72h. The investigators will then compare the rates of wound infection and wound complications between these two groups.

It is our hypothesis that negative pressure wound systems will decrease the wound infection and complication rate in this high risk population.

DETAILED DESCRIPTION:
Infectious complications have been found to be five times higher in women undergoing a cesarean delivery compared to a vaginal delivery. Known risk factors for wound complications are obesity, premature rupture of membranes, diabetes mellitus, hypertensive disorders, emergency cesarean delivery, twin delivery, chorioamnionitis, increased surgical blood loss and preeclampsia.

This study is aimed at determining whether or not the use of a suction device placed on the wound instead of a standard sterile dressing will decrease the prevalence of wound complications and wound infections in women at high risk for post operative complications. The investigators will compare the results from the participants of this study to an existing data set of historical controls who underwent cesarean delivery. The study involves placing a single use, portable negative wound pressure system kept in place while in the hospital after surgery (on average 48-72 hours) in women who meet criteria for increased risk of wound complications. The investigators will then compare the rates of wound infection and wound complications between these two groups.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* Having a cesarean delivery
* Has one or more of the following conditions:
* BMI > 30
* Anemia
* Preeclampsia (sever or mild)
* Hemolysis, elevated liver enzymes and low platelets (HELLP)
* Urgent procedure
* Rupture of membranes prior to surgery for > 4 hours
* Chorioamnionitis
* Hypertension
* Diabetes (Gestational or pre-gestational)
* Dense adhesive disease

Exclusion Criteria:

* Age < 18 years old
* Unable to give informed consent

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2012-08; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sara Tikkanen, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Negative Pressure Pump
Started | 110
Completed | 110
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Negative Pressure Pump
Number analyzed (Participants) | 110
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 110
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.8 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 110

OUTCOME MEASURES:

1. Primary Outcome: Wound Complication Rate
Description: Wound infection, separation or deep infection
Time Frame: Up to 6 weeks from time of surgery
Measure: Number; unit: participants
Arm/Group | Negative Pressure Pump
Number analyzed (Participants) | 110
participants
  wound infection | 3
  Endometritis | 1
  Wound separation | 3
  All wound complications (separation and infection) | 6

ADVERSE EVENTS:
Arm/Group | Negative Pressure Pump
All-Cause Mortality (participants affected / at risk) | 0/110
Serious Adverse Events (participants affected / at risk) | 1/110
Other Adverse Events (participants affected / at risk) | 0/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Negative Pressure Pump (N=110)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 — Skin irritation from negative pressure dressing

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No